CLINICAL TRIAL: NCT04651777
Title: Evaluation of Triple Therapy Using Magnetic Resonance Imaging in Asthma
Acronym: ETHA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. Grace Parraga (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor-Investigator, Dr. Grace Parraga, Professor, Western University, Canada
Organization: Western University, Canada (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ROB0046
Record Dates: First submitted 2020-11-19; First posted 2020-12-03 (Actual); Results first posted 2024-03-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Asthma
Keywords: Fluticasone furoate; umedlidinium; Vilanterol; Triple Therapy; Xenon
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: single arm, open-label pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants with poorly controlled moderate to severe asthma (Experimental): Participants with poorly controlled moderate to severe asthma will be evaluated during and after a six week trial of triple therapy (ICS/LABA/LAMA) for changes in 129Xe MRI ventilation percent defect, pulmonary function measurements.
  Interventions: Drug: FF/UMEC/VI

INTERVENTIONS:
Drug: FF/UMEC/VI — The investigational drug is a single Ellipta inhaler containing 200 ug fluticasone furoate, 62.5 ug umedlidinium and 25 ug vilanterol. The drug is delivered in an Ellipta inhaler in a single dose once daily.
  Other Names: Trelegy

SUMMARY:
The purpose of this study is to evaluate the effectiveness of treatment with triple therapy an inhaler that contains three types of asthma medications, on participants with poorly controlled asthma. The triple therapy medication contains fluticasone furoate, an inhaled corticosteroid (ICS) which reduces inflammation in the lungs; umeclidinium (UMEC), a long-acting muscarinic antagonist (LAMA), a medication which helps open up the airways; and vilanterol (VI), a long-acting beta2-adrenergic agonist (LABA) which also helps open up airways, delivered in a single daily inhalation via an Ellipta inhaler. The Investigators will evaluate lung structure and function using magnetic resonance imaging (MRI). Participants will inhale xenon gas before an MRI image of their lungs is taken. Using a special technique xenon is visible in MRI images, so this lets us see how air spreads in the lungs. In healthy lungs, the gas fills the lungs evenly, but in unhealthy lungs, the gas may fill the lungs unevenly and they will appear patchy. The patchy areas are called ventilation defects. A CT of the chest will be done to assess the structure of the lungs. The Investigators will also be using lung function testing and questionnaires to compare them to MRI ventilation defect measurements.

DETAILED DESCRIPTION:
This is an open-label, single arm pilot study in participants prescribed low or medium dose ICS/LABA inhaled therapy and poorly controlled asthma to quantify hyperpolarized 129Xe MRI VDP before and after six weeks of therapy with FF/UMEC/VI 200/62.5/25 ug QD. Male and females between 18 and 70 years of age will provide written informed consent to five visits including screening (Visit 1 week -2), baseline (Visit 2 week 0), mid-study Visit 3 in week 3, study end (Visit 4, week +6) and safety follow-up (Visit 5 week +8). The general study procedures are the same for Visit 1/Day -14, Visit 2/Day 0 and Visit 4/Day 42. Visit 3/Day 21 is an optional clinic visit or phone call. Visit 5 is a phone call check-in for adverse events.

For Visits 1, 2 and 4, participants are to withhold their medication as previously described. Vital signs will be recorded at the beginning of the visit. FeNO, spirometry, plethysmography, FOT, MBNW and 129Xe MRI will be performed pre-bronchodilator. FeNO will be performed before all other pulmonary function testing. Following 129Xe MRI, all participants will inhale 4 puffs (100mcg each) of a bronchodilator and quietly rest for 15 minutes. After 15 minutes, participants will undergo post-bronchodilator 129Xe MRI, and once MRI is complete, participants will undergo post-bronchodilator spirometry, plethysmography, FOT and MBNW. SGRQ, ACQ-6 and AQLQ will be administered after post-bronchodilator assessments are completed. For Visit 3, participants who choose to attend an in-person visit are to withhold their medication as described and the process for Visits 1, 2 and 4 will be followed. Participants who choose a phone call Visit 3 will be asked a series of questions regarding their breathing, asthma control and general health and they will complete the SGRQ, ACQ and AQLQ. For all participants, Visit 5 will entail a phone call check-in for adverse events. CT will be acquired at Visit 2, whilst MRI will be acquired on Visits 2, 4 and for those who prefer an in person visit, on Visit 3.

ELIGIBILITY:
Inclusion Criteria:

* Participant understands study procedures and is willing to participate in the study as indicated by the participant's signature
* Provision of written, informed consent prior to any study specific procedures
* Males and females with a clinical diagnosis of eosinophilic asthma (based on FENO ≥40ppb, blood eosinophilia≥ 200 cells/μl at screening) aged 18 to 70 years, inclusively, at the time of Visit 1 (enrolment), under the care of a respirologist
* FEV1 ≥35 and ≤80% predicted
* Participant is a current non-smoker and non-vaper, having not smoked tobacco or cannabis, pipe or cigar or vaped any product for at least 12 months prior to the study with a tobacco smoking history of no more than 1 pack-year (i.e. 1 pack per day for 1 year).
* Women of childbearing potential (after menarche) must use a highly effective form of birth control (confirmed by the investigator or designee)
* A highly effective form of birth control includes true sexual abstinence, a vasectomized sexual partner, Implanon®, female sterilization by tubal occlusion, any effective intrauterine device (IUD)/levonorgestrel intrauterine system (IUS), Depo-ProveraTM injections, oral contraceptive and Erva PatchTM or NuvaringTM
* Women of childbearing potential (after menarche) must agree to use a highly effective form of birth control, as defined above, from enrolment, throughout the study duration, and 8 weeks after last dose of study drug, with negative pregnancy test result at Visit 1
* Male participants who are sexually active must agree to use a double barrier method of contraception (condom with spermicide) from the first dose of the study drug until 8 weeks after last dose
* Participant has documented treatment with a stable dose of low to medium dose inhaled corticosteroids (defined as >250 and ≤500 mcg fluticasone proprionate/day or equivalent or, >400 to ≤800 mcg Budesonide/day for at least 6 months prior to enrolment
* long-acting β2-agonist (LABA) for at least 6 months prior to enrolment
* Participant has blood eosinophils ≥ 200 cells/μl or FENO ≥25ppb at Visit 1 for all participants except for those with previous biologic therapy without washout who will be required to washout prior to screening.
* Participant has ACQ-6 ≥ 1.5 at visit 1
* Participant has a history of poorly controlled asthma (i.e. ≥ 2 exacerbations in past 24 months)

Exclusion Criteria:

* Participant is, in the opinion of the investigator, mentally or legally incapacitated, preventing informed consent from being obtained, or cannot read or understand written material
* Participant has clinically important pulmonary disease other than asthma (e.g. active lung infection, chronic obstructive pulmonary disease, bronchiectasis, pulmonary fibrosis, cystic fibrosis, hypoventilation syndrome associated with obesity, lung cancer, alpha-1 antitrypsin deficiency and primary ciliary dyskinesia) or been diagnosed with pulmonary or systemic disease other than asthma that is associated with elevated peripheral eosinophil counts (e.g. allergic bronchopulmonary aspergillosis/mycosis, Churg-Strauss syndrome, hypereosinophilic syndrome), except for those atopic conditions that can be associated with asthma (e.g. allergic rhinitis, sinusitis with or without polyposis, eczema, and eosinophilic esophagitis)
* Any disorder, including, but not limited to, cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, haematological, psychiatric, or major physical impairment that is not stable in the opinion of the Qualified Investigator and/or could affect the safety of the participant throughout the study, influence the findings of the study or their interpretations, or impede the participant's ability to complete the entire duration of the study, as assessed by the Qualified Investigator.
* Known history of allergy or reaction to the study drug formulation
* Acute upper or lower respiratory infections requiring antibiotics or antiviral medication within 30 days prior to the date of informed consent
* Clinically significant asthma exacerbation, defined as a change from baseline deemed clinically relevant in the opinion of the Qualified investigator, including those requiring the use of OCS, or an increase in maintenance dosage of OCS within 30 days prior to the date of informed consent. Participants with an exacerbation after providing informed consent but prior to treatment start will be excluded from the study
* Receipt of immunoglobulin or blood products within 30 days prior to the date of informed consent
* Receipt of live attenuated vaccines 30 days prior to the date of enrolment
* Previously randomized in any FF/UMEC/VI 200/62.5/25ug study
* Planned surgical procedure during the conduct of the study
* Concurrent enrolment in another clinical trial
* Participant has history of alcohol or drug abuse within 12 months prior to the date of informed consent
* Participant is a female who is ≤8 weeks post-partum or breast feeding an infant
* Participant is pregnant, or intends to become pregnant during the time course of the study
* Participant is unable to perform MRI breath-hold maneuver
* Participant is unable to perform spirometry maneuver
* Participant is hospitalized or has had a major surgical procedure, major trauma requiring medical attention, or significant illness requiring medical attention within 4 weeks of Visit 1
* Participant has a blood pressure of >150 mmHg systolic or >95 mmHg diastolic on more than 2 measurements done >5 minutes apart at Visit 1
* In the opinion of the investigator, participant suffers from any physical, psychological or other condition(s) that might prevent performance of the MRI, such as severe claustrophobia
* Participant has implanted mechanically, electrically or magnetically activated device or any metal in their body, which cannot be removed, including but not limited to pacemakers, neurostimulators, biostimulators, implanted insulin pumps, aneurysm clips, bioprosthesis, artificial limb, metallic fragment or foreign body, shunt, surgical staples (including clips or metallic sutures and/or ear implants) - at the discretion of the MRI Technologist.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-08-08 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2025-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Grace E Parraga, PhD, Principal Investigator — Robarts Research Institute, The University of Western Ontario
Locations (1):
- Robarts Research Institute; The University of Western Ontario; London Health Sciences Centre, London, Ontario, Canada

REFERENCES:
- [Background] Kerwin E, Pascoe S, Bailes Z, Nathan R, Bernstein D, Dahl R, von Maltzahn R, Robbins K, Fowler A, Lee L. A phase IIb, randomised, parallel-group study: the efficacy, safety and tolerability of once-daily umeclidinium in patients with asthma receiving inhaled corticosteroids. Respir Res. 2020 Jun 12;21(1):148. doi: 10.1186/s12931-020-01400-5. PMID 32532275
- [Background] Global Initiative for Asthma (GINA). Global Strategy for Asthma Management and Prevention: Updated 2017. (2017).
- [Background] Dreher M, Muller T. Add-on Therapy for Symptomatic Asthma despite Long-Acting Beta-Agonists/Inhaled Corticosteroid. Tuberc Respir Dis (Seoul). 2018 Jan;81(1):1-5. doi: 10.4046/trd.2017.0102. Epub 2017 Dec 13. PMID 29256220
- [Background] Walford HH, Doherty TA. Diagnosis and management of eosinophilic asthma: a US perspective. J Asthma Allergy. 2014 Apr 11;7:53-65. doi: 10.2147/JAA.S39119. eCollection 2014. PMID 24748808
- [Background] de Groot JC, Ten Brinke A, Bel EH. Management of the patient with eosinophilic asthma: a new era begins. ERJ Open Res. 2015 Sep 23;1(1):00024-2015. doi: 10.1183/23120541.00024-2015. eCollection 2015 May. PMID 27730141
- [Background] Fain S, Schiebler ML, McCormack DG, Parraga G. Imaging of lung function using hyperpolarized helium-3 magnetic resonance imaging: Review of current and emerging translational methods and applications. J Magn Reson Imaging. 2010 Dec;32(6):1398-408. doi: 10.1002/jmri.22375. PMID 21105144
- [Background] Altes TA, Powers PL, Knight-Scott J, Rakes G, Platts-Mills TA, de Lange EE, Alford BA, Mugler JP 3rd, Brookeman JR. Hyperpolarized 3He MR lung ventilation imaging in asthmatics: preliminary findings. J Magn Reson Imaging. 2001 Mar;13(3):378-84. doi: 10.1002/jmri.1054. PMID 11241810
- [Background] Aysola R, de Lange EE, Castro M, Altes TA. Demonstration of the heterogeneous distribution of asthma in the lungs using CT and hyperpolarized helium-3 MRI. J Magn Reson Imaging. 2010 Dec;32(6):1379-87. doi: 10.1002/jmri.22388. PMID 21105142
- [Background] Svenningsen S, Kirby M, Starr D, Coxson HO, Paterson NA, McCormack DG, Parraga G. What are ventilation defects in asthma? Thorax. 2014 Jan;69(1):63-71. doi: 10.1136/thoraxjnl-2013-203711. Epub 2013 Aug 16. PMID 23956019
- [Background] Campana L, Kenyon J, Zhalehdoust-Sani S, Tzeng YS, Sun Y, Albert M, Lutchen KR. Probing airway conditions governing ventilation defects in asthma via hyperpolarized MRI image functional modeling. J Appl Physiol (1985). 2009 Apr;106(4):1293-300. doi: 10.1152/japplphysiol.91428.2008. Epub 2009 Feb 12. PMID 19213937
- [Background] Costella S, Kirby M, Maksym GN, McCormack DG, Paterson NA, Parraga G. Regional pulmonary response to a methacholine challenge using hyperpolarized (3)He magnetic resonance imaging. Respirology. 2012 Nov;17(8):1237-46. doi: 10.1111/j.1440-1843.2012.02250.x. PMID 22889229
- [Background] Kruger SJ, Niles DJ, Dardzinski B, Harman A, Jarjour NN, Ruddy M, Nagle SK, Francois CJ, Sorkness RL, Burton RM, Munoz del Rio A, Fain SB. Hyperpolarized Helium-3 MRI of exercise-induced bronchoconstriction during challenge and therapy. J Magn Reson Imaging. 2014 May;39(5):1230-7. doi: 10.1002/jmri.24272. Epub 2013 Sep 4. PMID 24006239
- [Background] Samee S, Altes T, Powers P, de Lange EE, Knight-Scott J, Rakes G, Mugler JP 3rd, Ciambotti JM, Alford BA, Brookeman JR, Platts-Mills TA. Imaging the lungs in asthmatic patients by using hyperpolarized helium-3 magnetic resonance: assessment of response to methacholine and exercise challenge. J Allergy Clin Immunol. 2003 Jun;111(6):1205-11. doi: 10.1067/mai.2003.1544. PMID 12789218
- [Background] Tzeng YS, Lutchen K, Albert M. The difference in ventilation heterogeneity between asthmatic and healthy subjects quantified using hyperpolarized 3He MRI. J Appl Physiol (1985). 2009 Mar;106(3):813-22. doi: 10.1152/japplphysiol.01133.2007. Epub 2008 Nov 20. PMID 19023025

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Participants With Poorly Controlled Moderate to Severe Asthma
Started | 31
Completed V1+V2 | 28
Completed | 28
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: All enrolled, Completed Visit 1
Arm/Group | Participants With Poorly Controlled Moderate to Severe Asthma
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 31
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index
  kg/m^2 | 31 (7)
Pre-BD FEV1 [Mean (Standard Deviation); unit: L] — Post Bronchodilator Forced Expiratory Volume in 1 second
  L | 2.1 (0.7)
Post-BD FEV1 [Mean (Standard Deviation); unit: L] — Pre Bronchodilator Forced Expiratory Volume in 1 second
  L | 2.4 (0.8)
Pre-BD Percentage of Predicted FEV1 [Mean (Standard Deviation); unit: percentage predicted] — Pre Bronchodilator Forced Expiratory Volume in 1 second
  percentage predicted | 72 (19)
Post-BD Percentage of Predicted FEV1 [Mean (Standard Deviation); unit: percentage predicted] — Post Bronchodilator Forced Expiratory Volume in 1 second
  percentage predicted | 81 (19)
Pre-BD FEV1/FVC [Mean (Standard Deviation); unit: percentage of FEV1/FVC] — Pre Bronchodilator Forced Expiratory Volume in 1 second/Forced Vital Capacity
  percentage of FEV1/FVC | 65 (12)
Post-BD FEV1/FVC [Mean (Standard Deviation); unit: percentage of FEV1/FVC] — Post Bronchodilator Forced Expiratory Volume in 1 second/Forced Vital Capacity
  percentage of FEV1/FVC | 68 (12)
Pre-BD RV/TLC [Mean (Standard Deviation); unit: percentage] — Pre Bronchodilator Residual Volume/Total Lung Capacity
  percentage | 44 (11)
Post-BD RV/TLC [Mean (Standard Deviation); unit: percentage] — Post Bronchodilator Residual Volume/Total Lung Capacity
  percentage | 37 (12)
Pre-BD Proximal Airway Resistance at 5 Hz (R5) [Mean (Standard Deviation); unit: cm H2O sec/L] | 5.7 (1.7)
Post-BD Proximal Airway Resistance at 5 Hz (R5) [Mean (Standard Deviation); unit: cm H2O sec/L] | 4.9 (1.5)
Pre-BD Proximal Airway Resistance at 19 Hz (R19) [Mean (Standard Deviation); unit: cm H2O sec/L] | 3.7 (1.2)
Post-BD Proximal Airway Resistance at 19 Hz (R19) [Mean (Standard Deviation); unit: cm H2O sec/L] | 3.5 (1.0)
Pre-BD Proximal Airway Resistance at 5 Hz -19Hz (R5-19) [Mean (Standard Deviation); unit: cm H2O sec/L] | 2.0 (1.0)
Post-BD Proximal Airway Resistance at 5 Hz - 19 Hz (R5-19) [Mean (Standard Deviation); unit: cm H2O sec/L] | 1.4 (0.9)
ACQ-6 [Mean (Standard Deviation); unit: units on a scale] — Asthma Control Questionnaire (ACQ-6) is used to evaluate asthma control. The ACQ-6 is scored from 0 to 6, with higher scores indicating more severely uncontrolled asthma.
  units on a scale | 2.0 (1.0)
AQLQ [Mean (Standard Deviation); unit: units on a scale] — Asthma Quality of Life Questionnaire with Standardised Activities (AQLQ(S)) evaluates asthma-related quality of life. The AQLQ(S) is scored from 1-7, with lower scores indicating more severe impairment.
  units on a scale | 4.5 (1.2)
SGRQ [Mean (Standard Deviation); unit: units] — The St. George's Respiratory Questionnaire (SGRQ) is a 2-part questionnaire with a score of 0-100, with higher numbers indicating more limitations.
  units | 49 (16)
Pre-BD VDP [Mean (Standard Deviation); unit: percentage] — Pre Bronchodilator Ventilation Defect Percent
  percentage | 15.5 (12.9)
Post-BD VDP [Mean (Standard Deviation); unit: percentage] — Post Bronchodilator Ventilation Defect Percent
  percentage | 10.7 (10.5)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Airway Function Measured Using 129-Xenon MRI Ventilation Defect Percent at the End of 6 Weeks of Treatment With FF/UMEC/VI 200/62.5/25ug Once Daily
Description: Change in VDP
Time Frame: Day 0 to day 42
Population: One participant did not complete imaging due to non-MR compatible pacemaker. One participant experienced claustrophobia and could not complete a scan at visit 2. Two participants' scans had technical errors which prevented VDP calculation.
Measure: Mean (Standard Deviation); unit: ventilation defect percent
Arm/Group | Participants With Poorly Controlled Moderate to Severe Asthma
Number analyzed (Participants) | 24
ventilation defect percent | 5 (12)

2. Secondary Outcome: Change From Baseline Forced Expiration Volume in One Second
Description: Indicator of pulmonary function
Time Frame: Baseline and Day 42
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Participants With Poorly Controlled Moderate to Severe Asthma
Number analyzed (Participants) | 28
L | 0.178 (0.516)

3. Secondary Outcome: Change From Baseline Forced Vital Capacity
Description: Indicator of pulmonary function
Time Frame: Baseline and Day 42
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Participants With Poorly Controlled Moderate to Severe Asthma
Number analyzed (Participants) | 28
L | 0.004 (0.634)

4. Secondary Outcome: Change From Baseline Residual Volume
Description: Indicator of pulmonary function
Time Frame: Baseline and Day 42
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Participants With Poorly Controlled Moderate to Severe Asthma
Number analyzed (Participants) | 28
L | 0.084 (1.88)

5. Secondary Outcome: Change From Baseline Total Lung Capacity
Description: Indicator of pulmonary function
Time Frame: Baseline and Day 42
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Participants With Poorly Controlled Moderate to Severe Asthma
Number analyzed (Participants) | 28
L | 0.385 (2.253)

6. Secondary Outcome: Change From Baseline in Proximal Airway Reactance at 5 Hz (R5), 19 Hz (R19), and 5 Hz - 19 Hz (R5-19)
Description: Indicator of pulmonary function and inflammation
Time Frame: Baseline and Day 42
Measure: Mean (Standard Deviation); unit: cm H2O sec/L
Arm/Group | Participants With Poorly Controlled Moderate to Severe Asthma
Number analyzed (Participants) | 28
cm H2O sec/L
  R5 | -1.1 (1.187)
  R19 | -0.36 (0.681)
  R5-19 | -0.737 (0.724)

7. Secondary Outcome: Change From Baseline Lung Clearance Index
Description: Lung clearance index is the number of breaths it takes until the exhaled nitrogen concentration is <2.5% of the concentration at the start of the test. It is an indicator of pulmonary function. A lower value is considered better as it indicates it takes a lower number of breaths for the nitrogen to exit the lungs.
Time Frame: Baseline and Day 42
Measure: Mean (Standard Deviation); unit: number of breaths
Arm/Group | Participants With Poorly Controlled Moderate to Severe Asthma
Number analyzed (Participants) | 28
number of breaths | -0.814 (4.045)

8. Secondary Outcome: Change From Baseline in Asthma Control
Description: Asthma Control Questionnaire (ACQ-6) is used to evaluate asthma control. The ACQ-6 is scored from 0 to 6, with higher scores indicating more severely uncontrolled asthma.
Time Frame: Baseline and Day 42
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants With Poorly Controlled Moderate to Severe Asthma
Number analyzed (Participants) | 28
score on a scale | -0.654 (1.333)

9. Secondary Outcome: Change From Baseline in Asthma-related Quality of Life
Description: Asthma Quality of Life Questionnaire with Standardised Activities (AQLQ(S)) evaluates asthma-related quality of life. The AQLQ(S) is scored from 1-7, with lower scores indicating more severe impairment.
Time Frame: Baseline and Day 42
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants With Poorly Controlled Moderate to Severe Asthma
Number analyzed (Participants) | 28
score on a scale | 0.862 (1.431)

10. Secondary Outcome: Change From Baseline in Daily Life and Perceived Well-being Using the SGRQ.
Description: The St. George's Respiratory Questionnaire (SGRQ) is a 2-part questionnaire with a score of 0-100, with higher numbers indicating more limitations.
Time Frame: Baseline and Day 42
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants With Poorly Controlled Moderate to Severe Asthma
Number analyzed (Participants) | 28
score on a scale | -12 (21)

ADVERSE EVENTS:
Time Frame: 9 Months
Arm/Group | Participants With Poorly Controlled Moderate to Severe Asthma
All-Cause Mortality (participants affected / at risk) | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 16/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Poorly Controlled Moderate to Severe Asthma (N=31)
Chest Infection (Infections and infestations) | 5
COVID-19 Infection (Infections and infestations) | 2
Light-headedness During Breath-hold (Nervous system disorders) | 2
Dry Mouth (General disorders) | 1
Gastroenteritis (Gastrointestinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Increased Nocturnal Awakening (Respiratory, thoracic and mediastinal disorders) | 1
Increased Mucous/Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 — Increased mucous/wheezing - ER admission
Rib Fracture (Respiratory, thoracic and mediastinal disorders) | 1 — Motor Vehicle Accident
Increased Appetite (Gastrointestinal disorders) | 1
Chest Congestion (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-08): https://cdn.clinicaltrials.gov/large-docs/77/NCT04651777/Prot_SAP_000.pdf